CLINICAL TRIAL: NCT04429971
Title: Pre-Exposure Prophylaxis Provision in the Emergency Department (PrEPPED): A Pilot Feasibility Study
Brief Title: Pre-Exposure Prophylaxis in the Emergency Department
Acronym: PrEPPED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Ethan Cowan, Director of Research and Community Engagement, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: GCO 19-2596
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: HIV/AIDS; PrEP
Keywords: Feasibility; Implementation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Part 1 of study will enroll 30 participants. Part 2 of study will enroll 40 participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immediate PreP initiation (Experimental): PreP screening program with immediate PrEP (iPrEP) initiation in the ED using a PrEP "starter pack" with facilitated linkage to care.
  Interventions: Other: PrEP screening program; Other: PrEP starter pack
- Out-patient care for PrEP initiation (Active Comparator): PrEP screening program with referral to out-patient care for PrEP initiation
  Interventions: Other: PrEP screening program
- PreP Screening Program (Experimental): Part 1: Targeted ED-based patients
  Interventions: Other: PrEP screening program

INTERVENTIONS:
Other: PrEP screening program — ICAP Pre-Exposure Prophylaxis (PrEP) Screening for Substantial Risk and Eligibility tool
Other: PrEP starter pack — emtricitabine/tenofovir alafenamide or emtricitabine/tenofovir disoproxil
  Arms: Immediate PreP initiation

SUMMARY:
Despite an increasing armamentarium of behavioral and biomedical HIV prevention methods, since 2010 rates of new infection have remained around 40,000 annually. The demonstrated efficacy and subsequent approval of emtricitabine/tenofovir disoproxil fumarate for pre-exposure prophylaxis (PrEP) for HIV by the FDA in 2012 was thought to represent a turning point that could significantly reduce the number of new infections. Since approval, the promise of PrEP as a transformative intervention has yet to be realized. Despite the implementation of systems for clinical evaluation for and initiation of PrEP by primary care providers, HIV specialists, and STI clinics, numerous barriers to PrEP expansion have been identified, including: 1) patient and provider lack of knowledge, 2) lack of access to medical care among high-risk individuals, 3) provider discomfort and inexperience with screening for risk behaviors, and 4) insurance and affordability. This proposal seeks to expand access to and engagement in PrEP among high risk individuals though an innovative delivery approach in the Emergency Department (ED) while addressing these four barriers.

DETAILED DESCRIPTION:
Aim 1: Initiate a targeted ED-based PrEP screening program and optimize its feasibility and acceptability.

1. Behavioral risk factor eligibility screening will be performed using the ICAP Pre-Exposure Prophylaxis (PrEP) Screening for Substantial Risk and Eligibility tool.
2. During a 3-month period, use continuous quality improvement methods to decrease the time for completion of PrEP eligibility screening to an interval that is acceptable to ED patients and providers.

Aim 2: Pre-Exposure Prophylaxis Provision in the ED (PrEPPED) Trial:

Identify 40 PrEP eligible patients over a 12-month period who are interested in initiating PrEP in the ED. These patients will be offered immediate PrEP (iPrEP) initiation in the ED with facilitated linkage to comprehensive out-patient care.

1. Evaluate the impact of a PrEP "starter pack" on patients agreeing to iPrEP. The primary outcome is engagement in care at 30-days post PrEP initiation visit. Secondary outcomes include retention in care, STI diagnosis, risk behavior and PrEP adherence.
2. Collect data on recruitment and attrition rates, as well as means and standard deviations for key measures that will be needed to plan a definitive trial of ED-initiated PrEP.

ELIGIBILITY:
Inclusion Criteria:

PrEP screen group:

* Patients 18 years of age and above
* Medically stable as determined by their provider
* Able to speak English
* Willing and able to consent to study participation.
* Not requiring hospital admission for ongoing care.

iPrep group:

* ED patients 18 years of age and above
* HIV negative determined by 4th generation rapid testing with no evidence of acute HIV infection as determined by their ED provider
* Medically stable as determined by their primary provider
* Able to speak English
* Able to consent to participation
* Contact information available for linkage
* Not requiring hospital admission for ongoing care.
* Eligible for PrEP based on CDC risk behavior and clinical criteria.

Exclusion Criteria:

PrEP screen group:

* ED patients younger than 18 years of age
* Medically or psychiatrically unstable as determined by the ED provider
* Unable to speak or understand English
* Unable to provide consent for study participation.
* Being admitted to the hospital for ongoing care

iPrEP group:

* ED patients younger than 18 years of age
* Known HIV positive or positive rapid HIV test in ED
* Medically or psychiatrically unstable as determined by the ED provider
* Unable to speak or understand English
* Unable to provide consent for study participation
* No means of re-contact upon ED discharge
* No behavioral risk factors indicating need for PrEP
* Medical contraindications to PrEP
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Cowan, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Beth Israel Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 1455 patients screened, 169 were eligible, 26 were randomized and received their assigned intervention.
Period: Overall Study
Arm/Group | Out-patient Care for PrEP Initiation | Immediate PreP Initiation
Started | 13 | 13
30-Day Completed | 9 | 10
60-Day Completed | 6 | 7
90-Day Completed | 6 | 5
Completed | 6 | 5
Not Completed | 7 | 8
Not completed — Lost to Follow-up | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Out-patient Care for PrEP Initiation | Immediate PreP Initiation | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29.0 [23 to 35] | 34 [28 to 39] | 32.5 [24 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 10 | 7 | 17
  Unknown or Not Reported | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black or African American | 4 | 8 | 12
  More than one race | 3 | 2 | 5
  White | 5 | 2 | 7
  Missing | 1 | 0 | 1
Highest level of education [Count of Participants; unit: Participants]
  Some high school, no diploma | 1 | 2 | 3
  High school graduate/GED or equivalent | 5 | 5 | 10
  Some college (4-year college or university) | 3 | 2 | 5
  College graduate (4-year college or university) | 3 | 3 | 6
  Post-college/graduate degree | 1 | 0 | 1
  Missing | 0 | 1 | 1
Estimated annual total income [Count of Participants; unit: Participants]
  < $1000 | 1 | 2 | 3
  $1001-$2500 | 0 | 1 | 1
  $5001-$10,000 | 1 | 0 | 1
  $10,001-$20,000 | 1 | 1 | 2
  $20,001-$40,000 | 0 | 3 | 3
  $40,001 or more | 5 | 4 | 9
  Don't know | 3 | 2 | 5
  Missing | 2 | 0 | 2
Past-year employment status [Count of Participants; unit: Participants]
  Disabled | 2 | 1 | 3
  Looking for work/unemployed | 3 | 3 | 6
  Student | 0 | 1 | 1
  Working full time | 5 | 4 | 9
  Working part time | 2 | 4 | 6
  Prefer not to answer | 1 | 0 | 1
Covered by health insurance/health plan [Count of Participants; unit: Participants] | 12 | 12 | 24
Frequency of having run out of money for basic necessities in the past year [Count of Participants; unit: Participants]
  Daily | 0 | 2 | 2
  Monthly | 1 | 1 | 2
  Never | 6 | 6 | 12
  Occasionally | 3 | 2 | 5
  Prefer not to answer | 1 | 0 | 1
  Weekly | 2 | 2 | 4
Experiencing homelessness [Count of Participants; unit: Participants]
  No | 13 | 10 | 23
  Yes | 0 | 3 | 3
Current living situation [Count of Participants; unit: Participants]
  In a rooming, boarding, or halfway house | 0 | 1 | 1
  On the street(s) (Vacant lot, abandoned building, park, etc.) | 0 | 1 | 1
  Other | 0 | 1 | 1
  Own or rent home/apartment | 12 | 7 | 19
  Shelter | 1 | 2 | 3
  Staying at home of friend(s)/other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Engagement in Care (Implementation Component)
Description: Engagement is care is defined by attending at least 1 out-patient clinic appointment with a PrEP provider within 30-days of the ED visit.
Time Frame: 30 days post-ED visit
Measure: Count of Participants; unit: Participants
Arm/Group | Out-patient Care for PrEP Initiation | Immediate PreP Initiation
Number analyzed (Participants) | 9 | 10
Participants | 1 | 1

2. Primary Outcome: Number of Participants on PrEP Usage
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Out-patient Care for PrEP Initiation | Immediate PreP Initiation
Number analyzed (Participants) | 6 | 5
Participants | 1 | 2

3. Secondary Outcome: PrEPPED Satisfaction and Acceptability Survey (RCT Component)
Description: PrEPPED Satisfaction and Acceptability Survey is a patient satisfaction questionnaire was developed by the study team. It's a series of independent Likert questions from 1-6 addressing different aspects of the program. Full scale from 0 to 18, with higher score indicating more satisfaction.
  Satisfaction data were not collected at 30, 60, or 90 days. After study initiation, it was determined by the researchers that the satisfaction items were specific to the emergency department visit experience and not relevant to the follow-up period. Consequently, decision was made to not administer the follow-up satisfaction assessments, therefore, no data was collected so there is no data to report.
Time Frame: 30 days post-ED visit
Population: No protocol amendment was generated for this Outcome Measure. Although the outcome was prespecified in the initial protocol, the study team ultimately determined during implementation that the required data elements could not be collected reliably across sites. Because this decision did not alter the study intervention, eligibility criteria, procedures, or primary outcome, and because no participant-facing activities were affected, the team did not submit a formal protocol amendment at the time.
Arm/Group | Out-patient Care for PrEP Initiation | Immediate PreP Initiation
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: The VSQ-9 is a Visit-specific Satisfaction Instrument (RCT Component)
Description: The VSQ-9 is a visit-specific satisfaction instrument adapted by the American Medical Guidelines Regimen Information Program (GRIP) survey. GRIP guide is a self-report to assess PrEP adherence at 30-days post ED visit, with 6 categorical items: excellent, very good, good, fair, poor, and very poor.
  Because participants were not required to follow up at a single clinic, post-discharge care settings varied widely. The VSQ-9 assesses satisfaction with a specific clinical encounter, and applying it across multiple, non-standardized settings was deemed inappropriate and unlikely to yield interpretable data. Therefore, decision was made by the researcher to not administer the VSQ-9 at 30, 60, or 90 days. Consequently, no follow-up VSQ-9 data were collected so there is no data to report.
Time Frame: 30 days post-ED visit
Population: as for outcome 3
Arm/Group | Out-patient Care for PrEP Initiation | Immediate PreP Initiation
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: CDC Sexual Behavior Questions (CSBQ) (RCT Component)
Description: CDC Sexual Behavior Questions (CSBQ) to measure HIV risk behavior. CSBQ is a multi-tiered, gender-specific questionnaire developed by the Centers for Disease Control and Prevention HIV-STID Behavioral Surveillance Working Group. Three separate domains - Sexual Behavior, Drug-related HIV risk, and HIV testing. Responses are yes/no with no summation.
  Number of participants who engaged in unsafe sexual behavior, was under substance influence and who had a HIV test.
Time Frame: 30 days post-ED visit
Measure: Count of Participants; unit: Participants
Arm/Group | Out-patient Care for PrEP Initiation | Immediate PreP Initiation
Number analyzed (Participants) | 9 | 10
Participants
  Sexual Behavior | 4 | 5
  Drug-related HIV risk | 2 | 2
  HIV testing | 0 | 0

6. Secondary Outcome: Number of Participants of New STI Diagnoses (RCT Component)
Description: Number of new STI diagnosis between day 1 (day after enrollment) and day 90 (final day of follow-up) broken down into days 1-30, 31-60, 61-90.
Time Frame: 30 days, 60 days, and 90 days post-ED visit
Population: Number of new STI diagnosis between day 1 (day after enrollment) and day 90 (final day of follow-up) broken down into days 1-30, 31-60, 61-90. Number analyzed at each time differ due to participants being lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Out-patient Care for PrEP Initiation | Immediate PreP Initiation
Number analyzed (Participants) | 9 | 10
Participants
  day 1 to day 30 | 1 | 2
  day 31 to day 60: number analyzed (Participants) | 6 | 7
  day 31 to day 60 | 0 | 0
  day 61 to day 90: number analyzed (Participants) | 6 | 5
  day 61 to day 90 | 0 | 0

7. Secondary Outcome: Number of Participants of New HIV Infection (RCT Component)
Description: Number of new HIV diagnosis at 90-days after enrollment. This question was only asked for those individuals who had not been lost to follow-up.
Time Frame: 90 days post-ED visit
Population: Number of new HIV diagnosis at 90-days after enrollment. This question was only asked for those individuals who had not been lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Out-patient Care for PrEP Initiation | Immediate PreP Initiation
Number analyzed (Participants) | 6 | 5
Participants | 0 | 0

ADVERSE EVENTS:
Description: not collected
Arm/Group | Out-patient Care for PrEP Initiation | Immediate PreP Initiation
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT04429971/Prot_SAP_000.pdf